Version 1 – 03/12/18 IRAS ID:



## **CONSENT FORM**

Does pregnancy induce changes in Urinary C-peptide Creatinine Ratio (UCPCR) in women with Type 1 diabetes?

| 1. | I have been given the opportunity to ask questions and discuss the study | |
|---|---|---|
| 2. | I have received satisfactory answers to all my questions | |
| 3. | I have received enough information about the study | |
| 4. | I confirm that I have read and understand the information sheet dated, version "Does pregnancy induce changes in Urinary C-peptide Creatinine Ratio (UCPCR) in women Type 1 diabetes?." for the above study. | |
| 5. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | |
| 6. | I understand that sections of any of my medical notes/records may be looked at by responsible individuals from Imperial College NHS Healthcare Trust and regulatory authorities where it is relevant to my taking part in research. I give permission for these individuals to have access to my records. | |
| 7. | I understand that the data collected for this study will be securely stored at Imperial College NHS Trust for 10 years following completion of the study. | |
| 8. | I authorise this consent form to be store in the study's Master file at Imperial College London NHS Trust. | |
| 9. | I authorise the research team to use data previously collected from the booking visit for the purposes of this study. | |
| 10. | I authorise the research team to inform my GP that I will be taking part in this study. | |
| 11. | I agree to have placental tissue samples collected to collaborate with the Beta cell neogenesis research. Yes N | 0 |

| 12. | I to take part in this study. | | |
|-----|--------------------------------------------|-----------|-----------|
| 13. | I would like to be contacted regarding the | Yes No | |
| Nam | ne of Patient | Date | Signature |
| Res | earcher | Signature | Date |

1 for patient; 1 for researcher; 1 to be kept with hospital notes